CLINICAL TRIAL: NCT03101865
Title: An Open-label, Multi-centre, Randomised, 2-period Cross-over Study to Assess the Efficacy and Safety of Closed Loop Insulin Delivery Using Diluted Insulin in Comparison With Closed Loop With Non-diluted Insulin Over 21 Days in Children With Type 1 Diabetes Aged 1 to 7 Years in the Home Setting
Brief Title: The Artificial Pancreas in Very Young Children With T1D - Pilot (KidsAP01)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: European Commission (Other); Medtronic (Industry); Cambridge University Hospitals NHS Foundation Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); University of Luxembourg (Other); University of Leipzig (Other); Medical University of Graz (Other); Medical University Innsbruck (Other); Medical University of Vienna (Other); Jaeb Center for Health Research (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Director of Research, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: KidsAP01
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes; Artificial Pancreas; Closed-loop glucose control; Very young children; Continuous subcutaneous insulin infusion; Continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed loop with diluted insulin (Experimental): Unsupervised home use of day and night automated closed loop insulin delivery system (FlorenceM) combined with pump suspend feature using DILUTED insulin aspart over 3 weeks.
  Interventions: Device: FlorenceM
- Closed loop with standard insulin strength (Active Comparator): Unsupervised home use of day and night automated closed loop insulin delivery system (FlorenceM) combined with pump suspend feature using STANDARD strength insulin aspart over 3 weeks.
  Interventions: Device: FlorenceM

INTERVENTIONS:
Device: FlorenceM — The automated closed loop system (FlorenceM) will consist of: Next generation sensor augmented Medtronic insulin pump 640G (Medtronic Minimed, CA, USA) incorporating the Medtronic Enlite 3 family real time CGM and glucose suspend feature. An Android smartphone containing the Cambridge model predictive algorithm and communicating wirelessly with the insulin pump using a proprietary translator device.

SUMMARY:
The suggested clinical trial is part of the KidsAP project funded by the European Commission's Horizon 2020 Framework Programme. The project evaluates the use of the Artificial Pancreas (or closed loop systems) in very young children with type 1 diabetes (T1D) aged 1 to 7 years. The suggested trial is a feasibility study to pilot the setup of a large-scale outcome trial and to address the specific needs of this population. The results of the pilot trial will feed into the design of the outcome study.

In this study the investigators will compare closed loop insulin delivery using standard strength insulin to closed loop use with diluted insulin in very young children with T1D. Diluted insulin is a standard treatment approach for children with low insulin requirements. The investigators hypothesize that diluted insulin will lead to more stable glucose levels by reducing inaccuracies accentuated by delivery of minute amounts of insulin (frequently less than 0.1U/h [1μl/h with standard strength insulin] in small children compared to 1U/h in adults). These inaccuracies may result from pump plunger micro-jumps, tissues pressure build-up, and infusion set kinking. This study builds on previous and on-going studies of closed loop systems that have been performed in Cambridge in children and adolescents with T1D in clinical research facilities and in the home setting.

The study adopts an open-label, multi-centre, multinational, randomised, two-period crossover design contrasting closed loop glucose control using diluted insulin and closed loop using standard insulin strength under free-living home conditions. The two intervention periods will last 3 weeks each with a 1 to 4 weeks washout period in between. The order of the two interventions will be random. A total of up to 30 young children aged 1 to 7 years with T1D on insulin pump therapy will be recruited through outpatient diabetes clinics at participating clinical centres to allow for 24 completed subjects available for assessment in each of the study arms.

Prior to the use of study devices, participants and parents/guardians will receive appropriate training by the research team on the safe use of the study pump and continuous glucose monitoring system, and the hybrid closed loop insulin delivery system. Carers at nursery or school may also receive training by the study team if required. During the intervention periods, subjects and parents/guardians will use the closed loop system for 21 days under free-living conditions in their home and nursery/school environment without remote monitoring or supervision by research staff.

The primary outcome is time spent in target range between 3.9 and 10.0 mmol/l as recorded by CGM. Secondary outcomes are the time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics. Safety evaluation comprises the tabulation of severe hypoglycaemic episodes.

DETAILED DESCRIPTION:
Purpose of clinical trial:

This is a feasibility study to pilot the outcome study setup and to address the specific needs of the studied population by comparing closed loop insulin delivery using standard strength insulin (U-100) and diluted insulin. The results will feed into the design of a follow up outcome study. The investigators hypothesize that diluted insulin will lead to more stable glucose levels by reducing inaccuracies accentuated by delivery of small amounts of insulin (frequently less than 0.1U/h [1μl/h with standard strength insulin] in small children.

Study objectives:

The study objective is to evaluate the safety, efficacy and utility of day-and-night closed loop glucose control in young children with type 1 diabetes.

1. EFFICACY: The objective is to assess the ability of a day-and-night hybrid closed loop system using diluted insulin to maintain CGM glucose levels within the target range of 3.9 to 10mmol/l (70 to 180mg/dl) in comparison with a hybrid closed loop system with standard insulin strength in young children with type 1 diabetes.
2. SAFETY: The objective is to evaluate the safety of day-and-night closed loop using diluted insulin versus closed loop with non-diluted insulin in terms of episodes and severity of hypoglycaemia, and nature and severity of other adverse events.
3. UTILITY: The objective is to determine the overall acceptability and duration of use of the closed loop system in this population.

Study Design:

The pilot study adopts an open-label, multi-centre, multinational, randomised, two-period crossover study design contrasting closed loop glucose control using diluted insulin and closed loop using standard insulin strength in young children with type 1 diabetes in the home setting. Two intervention periods will last 3 weeks each with 1 to 4 weeks washout period. The order of the two interventions will be random.

Participating clinical centres:

1. Addenbrooke's Hospital, Cambridge University Hospital NHS Foundation Trust, Cambridge, UK
2. Leeds Teaching Hospitals NHS Trust, Leeds, UK
3. University of Luxembourg, Luxembourg
4. University of Leipzig, Leipzig, Germany
5. Medical University of Graz, Graz, Austria
6. Medical University of Innsbruck, Innsbruck, Austria
7. Medical University of Vienna, Vienna, Austria

Sample Size:

24 participants randomised (2-5 participants per centre), equal proportion of those with total daily insulin dose ≤12 U/day and >12 U/day

Maximum duration of study for a subject: 14 weeks

Recruitment:

The subjects will be recruited through paediatric diabetes outpatient clinics at participating clinical centres (see above). Enrollment will target up to 30 (2-5 participants per centre) to allow for dropouts during run-in (approximately equal proportion of those with total daily insulin dose ≤12 U/day and >12 U/day).

Consent:

Written informed consent will be obtained from all parents/guardians and written assent from older children before any study related activities.

Baseline Assessment:

Eligible subjects will undergo a baseline evaluation including a blood sample for the measurement of HbA1c. Questionnaires will be completed by parents/guardians.

Pre-Study Training and Run-in:

Training sessions on the use of the study CGM and insulin pump will be provided by the research team. During a 2-4 week run-in period, subjects will use study CGM and insulin pump. For compliance and to assess the ability of the subject to use the study devices safely, at least 8 days of CGM data need to be recorded and safe use of study insulin pump demonstrated during the last 14 days of run-in period. The CGM data will also be used to assess baseline glucose control and may be used for treatment optimization as necessary.

Competency Assessment:

Competency on the use of study insulin pump and study CGM will be evaluated using a competency assessment tool developed by the research team. Training may be repeated if required.

Randomisation:

Eligible subjects will be randomised to the use of automated hybrid closed loop glucose system with diluted insulin or to closed loop with standard strength insulin for 21 days, with a 1-4 week washout period in between the two interventions.

1. Closed loop with diluted insulin Training on the use of the closed loop system with diluted insulin will be provided by the research team. During this 2-4 hour session, subjects and parents/guardians will operate the system under the supervision of the clinical research team, practicalities around the use of diluted insulin will be discussed, and pump settings will be adjusted accordingly. Competency on the use of closed loop system will be evaluated. Thereafter, subjects and their parents/guardians will continue using the hybrid closed loop system with diluted insulin over 21 days at home.
2. Closed loop with standard insulin strength:

Identical procedures as described above will be followed including training on the use of the closed loop system with standard strength insulin. Subjects will continue using the closed loop system with standard strength insulin at home over 21 days.

End of study assessments:

Study devices will be downloaded and returned. Participants will resume usual care using their pre-study insulin pump. A closed loop experience questionnaire will be completed by parents/guardians.

Procedures for safety monitoring during trial:

Standard operating procedures for monitoring and reporting of all adverse events will be in place, including serious adverse events (SAE) and specific adverse events (AE) such as severe hypoglycaemia.

Criteria for withdrawal of subjects on safety grounds:

A subject/guardian may terminate participation in the study at any time without necessarily giving a reason and without any personal disadvantage. An investigator can stop the participation of a subject after consideration of the benefit/risk ratio. Possible reasons are:

* Serious adverse events
* Non-compliance
* Serious protocol violation
* Decision by the investigator, or the sponsor, that termination is in the subject's best medical interest

ELIGIBILITY:
Inclusion Criteria:

1. Age between 1 and 7 years of age (inclusive)
2. Type 1 diabetes as defined by WHO for at least 6 months
3. Insulin pump user (with or without continuous glucose monitoring or flash glucose monitoring system) for at least 3 months, with subject/carer good knowledge of insulin self-adjustment as judged by the investigator
4. Treated with rapid acting insulin analogue insulin Aspart (Novo Nordisk, Bagsvaerd, Denmark)
5. Subject/carer is willing to perform regular finger-prick blood glucose monitoring, with at least 4 blood glucose measurements taken every day
6. Screening HbA1c ≤ 11% (97mmol/mol)
7. Willing to wear glucose sensor
8. Willing to wear closed loop system 24/7
9. The subject/carer is willing to follow study specific instructions
10. The subject/carer is willing to upload pump and CGM data at regular intervals

Exclusion Criteria:

1. Physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
2. Untreated coeliac disease or thyroid disease based on local investigations prior to study enrolment
3. Current treatment with drugs known to interfere with glucose metabolism, e.g. systemic corticosteroids
4. Known or suspected allergy to insulin
5. Recurrent incidents of severe hypoglycaemia (>2 episodes) during the previous 6 months [severe hypoglycaemia is defined as an event associated with a seizure or loss of consciousness]
6. Unwilling to avoid regular use of acetaminophen
7. Carer's lack of reliable telephone facility for contact
8. Total daily insulin dose ≥ 2 IU/kg/day
9. Subject/carer's severe visual impairment
10. Subject/carer's severe hearing impairment
11. Medically documented allergy towards the adhesive (glue) of plasters or subject is unable to tolerate tape adhesive in the area of sensor placement
12. Serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) located in parts of the body which could potentially be used for localisation of the glucose sensor)
13. Sickle cell disease, haemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
14. Plan to receive red blood cell transfusion or erythropoietin over the course of study participation
15. Subject/carer not proficient in English (UK) or German (Germany, Austria, Luxembourg) or French (Luxembourg)

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Time in target (3.9 to 10.0mmol/l) (70 to 180 mg/dl) | 3-week home stay
  Percentage of time spent with sensor glucose readings in the target glucose range from 3.9 to 10.0 mmol// (70 to 180 mg/dl)

SECONDARY OUTCOMES:
Time spent below target glucose (3.9mmol/l)(70mg/dl) | 3-week home stay
  Percentage of time spent with sensor glucose readings below target glucose (3.9mmol/l)(70mg/dl)
Time spent above target glucose (10.0mmol/l) (180mg/dl) | 3-week home stay
  Percentage of time spent with sensor glucose readings above target glucose (10.0mmol/l) (180mg/dl)
Average glucose | 3-week home stay
  Average of sensor glucose levels
Standard deviation of glucose levels | 3-week home stay
  Standard deviation of sensor glucose levels
Coefficient of variation of glucose levels | 3-week home stay
  Coefficient of variation of sensor glucose levels
Time with glucose levels < 3.5mmol/l (63 mg/dl) | 3-week home stay
  Percentage of time spent with glucose levels < 3.5mmol/l (63 mg/dl)
Time with glucose levels <2.8mmol/l (50mg/dl) | 3-week home stay
  Percentage of time spent with glucose levels <2.8mmol/l (50mg/dl)
Time with glucose levels in significant hyperglycaemia | 3-week home stay
  Percentage of time spent with glucose levels in significant hyperglycaemia (glucose levels > 16.7mmol/l) (300mg/dl)
Total daily insulin dose | 3-week home stay
  Average total daily insulin requirements
Daily basal insulin dose | 3-week home stay
  Average daily basal insulin requirements
Daily bolus insulin dose | 3-week home stay
  Average daily bolus insulin requirements
AUC of glucose below 3.5mmol/l (63mg/dl) | 3-week home stay
  Area under the curve of sensor glucose readings below 3.5mmol/l (63mg/dl)

OTHER OUTCOMES:
Number of episodes of severe hypoglycaemia | 3-week home stay
  Safety evaluation
Number of subjects experiencing severe hypoglycaemia | 3-week home stay
  Safety evaluation
Frequency of diabetic ketoacidosis | 3-week home stay
  Safety evaluation
Frequency and nature of other adverse events or serious adverse events | 3-week home stay
  Safety evaluation
Percentage of time of closed-loop operations | 3-week home stay
  Utility evaluation
Percentage of time of CGM availability | 3-week home stay
  Utility evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Study Director — Department of Paediatrics, University of Cambridge, UK; Carlo Acerini, MD, Principal Investigator — Department of Paediatrics, University of Cambridge, UK; Carine de Beaufort, PhD, Principal Investigator — Clinique Pédiatrique de Luxembourg, University of Luxembourg, Luxembourg; Fiona Campbell, MD, Principal Investigator — St James's University Hospital, Leeds, UK; Elke Fröhlich-Reiterer, MD, Principal Investigator — Department of Pediatrics and Adolescent Medicine, Medical University of Graz, Graz, Austria; Sabine Hofer, MD, Principal Investigator — Department of Pediatrics I, Medical University of Innsbruck, Innsbruck, Austria; Thomas Kapellen, MD, Principal Investigator — Division for Paediatric Diabetology, University of Leipzig, Leipzig, Germany; Birgit Rami-Merhar, MD, Principal Investigator — Deptartment of Pediatrics, Medical University of Vienna, Vienna, Austria
Locations (7):
- Austria (3):
  - Department of Pediatrics and Adolescent Medicine, Medical University of Graz, Graz
  - Department of Pediatrics I, Medical University of Innsbruck, Innsbruck
  - Deptartment of Pediatrics, Medical University of Vienna, Vienna
- Division for Paediatric Diabetology, University of Leipzig, Leipzig, Germany
- Clinique Pédiatrique de Luxembourg, Luxembourg, Luxembourg
- United Kingdom (2):
  - University of Cambridge, Cambridge
  - St James's University Hospital, Leeds

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised data may be shared with third parties (EU or non-EU based) for the purposes of advancing management and treatment of diabetes.

REFERENCES:
- [Background] Elleri D, Allen JM, Tauschmann M, El-Khairi R, Benitez-Aguirre P, Acerini CL, Dunger DB, Hovorka R. Feasibility of overnight closed-loop therapy in young children with type 1 diabetes aged 3-6 years: comparison between diluted and standard insulin strength. BMJ Open Diabetes Res Care. 2014 Dec 11;2(1):e000040. doi: 10.1136/bmjdrc-2014-000040. eCollection 2014. PMID 25512874
- [Background] Ruan Y, Elleri D, Allen JM, Tauschmann M, Wilinska ME, Dunger DB, Hovorka R. Pharmacokinetics of diluted (U20) insulin aspart compared with standard (U100) in children aged 3-6 years with type 1 diabetes during closed-loop insulin delivery: a randomised clinical trial. Diabetologia. 2015 Apr;58(4):687-90. doi: 10.1007/s00125-014-3483-6. Epub 2014 Dec 24. PMID 25537835
- [Background] Thabit H, Tauschmann M, Allen JM, Leelarathna L, Hartnell S, Wilinska ME, Acerini CL, Dellweg S, Benesch C, Heinemann L, Mader JK, Holzer M, Kojzar H, Exall J, Yong J, Pichierri J, Barnard KD, Kollman C, Cheng P, Hindmarsh PC, Campbell FM, Arnolds S, Pieber TR, Evans ML, Dunger DB, Hovorka R. Home Use of an Artificial Beta Cell in Type 1 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2129-2140. doi: 10.1056/NEJMoa1509351. Epub 2015 Sep 17. PMID 26379095
- [Background] Tauschmann M, Allen JM, Wilinska ME, Thabit H, Stewart Z, Cheng P, Kollman C, Acerini CL, Dunger DB, Hovorka R. Day-and-Night Hybrid Closed-Loop Insulin Delivery in Adolescents With Type 1 Diabetes: A Free-Living, Randomized Clinical Trial. Diabetes Care. 2016 Jul;39(7):1168-74. doi: 10.2337/dc15-2078. Epub 2016 Jan 6. PMID 26740634
- [Background] Tauschmann M, Allen JM, Wilinska ME, Thabit H, Acerini CL, Dunger DB, Hovorka R. Home Use of Day-and-Night Hybrid Closed-Loop Insulin Delivery in Suboptimally Controlled Adolescents With Type 1 Diabetes: A 3-Week, Free-Living, Randomized Crossover Trial. Diabetes Care. 2016 Nov;39(11):2019-2025. doi: 10.2337/dc16-1094. Epub 2016 Sep 9. PMID 27612500
- [Derived] Tauschmann M, Allen JM, Nagl K, Fritsch M, Yong J, Metcalfe E, Schaeffer D, Fichelle M, Schierloh U, Thiele AG, Abt D, Kojzar H, Mader JK, Slegtenhorst S, Barber N, Wilinska ME, Boughton C, Musolino G, Sibayan J, Cohen N, Kollman C, Hofer SE, Frohlich-Reiterer E, Kapellen TM, Acerini CL, de Beaufort C, Campbell F, Rami-Merhar B, Hovorka R; KidsAP Consortium. Home Use of Day-and-Night Hybrid Closed-Loop Insulin Delivery in Very Young Children: A Multicenter, 3-Week, Randomized Trial. Diabetes Care. 2019 Apr;42(4):594-600. doi: 10.2337/dc18-1881. Epub 2019 Jan 28. PMID 30692242